CLINICAL TRIAL: NCT04597060
Title: The Safety and Efficacy of Thermo-mechanical System for Fractional Ablation Associated Triamcinolone Acetonide Drug Delivery for the Treatment of Hypertrophic Scars and Keloids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Si 719/2018
Record Dates: First submitted 2020-09-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Keloid
Keywords: Keloid, thermo-mechanical system
MeSH Terms: conditions — Keloid | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split Keloid - first side (Experimental)
  Interventions: Device: Thermomechanical system with corticosteroids
- Split Keloid - second side (Experimental)
  Interventions: Other: corticosteroid injection

INTERVENTIONS:
Device: Thermomechanical system with corticosteroids — The device in this study using Novoxel - Tixel®
  Arms: Split Keloid - first side
Other: corticosteroid injection — corticosteroid injection using TA 10mg/ml
  Arms: Split Keloid - second side

SUMMARY:
This study aims to assess the safety and efficacy of Thermo-mechanical system for fractional ablation associated triamcinolone acetonide drug delivery for the treatment of Hypertrophic scars and Keloids.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without underlying disease
* Patient with keloid age more than 6 months and keloid thickness more than 1 mm.

Exclusion Criteria:

* Dermatitis or infection on treatment area
* Suspected cancer on treatment area
* Immunocompromised host
* Pregnancy or lactating woman
* Recieved corticosteroid injection within 2 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Thickness by caliper (mm) - comparing between Thermo-mechanical system for fractional ablation associated triamcinolone acetonide drug delivery and triamcinolone acetonide injection for the treatment of Hypertrophic scars and Keloids | 6 months
  cthickness by caliper in mm.
Vancouver Scar Scale - comparing between Thermo-mechanical system for fractional ablation associated triamcinolone acetonide drug delivery and triamcinolone acetonide injection for the treatment of Hypertrophic scars and Keloids | 6 months
  Vancouver Scar Scale between 0 to 13
Antera Elevation Volume - comparing between Thermo-mechanical system for fractional ablation associated triamcinolone acetonide drug delivery and triamcinolone acetonide injection for the treatment of Hypertrophic scars and Keloids | 6 months
  Measuring Antera Elevation Volume in mm3
Patient satisfaction quartile scale - comparing between Thermo-mechanical system for fractional ablation associated triamcinolone acetonide drug delivery and triamcinolone acetonide injection for the treatment of Hypertrophic scars and Keloids | 6 months
  Patient satisfaction quartile scale from 0 - 100%
Physician evaluation quartile score - comparing between Thermo-mechanical system for fractional ablation associated triamcinolone acetonide drug delivery and triamcinolone acetonide injection for the treatment of Hypertrophic scars and Keloids | 6 months
  Physician evaluation quartile score from 0-100%

SECONDARY OUTCOMES:
Side effect of Thermo-mechanical system, Triamcinolone itself, Injection side effect | 6 months
Side effect of Triamcinolone acetonide injection | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No